CLINICAL TRIAL: NCT01394081
Title: Alabama Veterans Rural Health Initiative
Acronym: AVRHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: Tuscaloosa Veterans Affairs Medical Center (U.S. Federal Agency); VA Office of Research and Development (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lori Davis, MD, ACOS Research and Development, Tuscaloosa Research & Education Advancement Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 00134
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2017-09

CONDITIONS: Problems With Access to Health Care; Health Behavior
Keywords: Veterans; Health Care Utilization; Rural Health; Patient Navigation; Motivational Interviewing
MeSH Terms: conditions — Health Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Prospective randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Engagement and Enrollment (EEE) (Experimental): Enhanced Engagement and Enrollment (EEE) consists of the outreach worker (interventionalist) engaging the participant in education (about VA resources and medical care), navigating the patient through the VA eligibility, enrollment, and scheduling processes, and using motivational interview to focus on ambivalence about attending a VA appointment.
  Interventions: Other: Enhanced Engagement and Enrollment (EEE)
- Administrative Outreach (AO) (Active Comparator): Administrative Outreach (AO) consists of the outreach worker giving the participants an application package to VA enrollment or phone number for the scheduling clerk. This intervention does not involve education, patient navigation (guidance through VA eligibility, enrollment, and scheduling processes) or motivational interviews (interviews focused on ambivalence about attending a VA appointment).
  Interventions: Other: Administrative Outreach (AO)

INTERVENTIONS:
Other: Enhanced Engagement and Enrollment (EEE) — Consists of motivational interviewing, educational outreach, and patient navigation.
  Other Names: Enhanced Engagement and Enrollment
  Arms: Enhanced Engagement and Enrollment (EEE)
Other: Administrative Outreach (AO) — Consists of giving information about enrolling for VA medical care or scheduling an appointment
  Other Names: Treatment-as-usual
  Arms: Administrative Outreach (AO)

SUMMARY:
The purpose of the Alabama Veterans Rural Health Initiative is to better understand access and barriers to health care and to enhance veteran enrollment or engagement in health care services of veterans residing in rural areas. It describes an intervention that is adaptable for use by other VA facilities that serve veterans in rural settings, and importantly, this study will improve our understanding of barriers to care and evaluate a method for enhancing access to care. The anticipated impact is that more veterans in rural areas who were previously under-utilizing VA services will receive and attend a health care appointment. This gain may improve preventative and primary care health care and reduce long term health care morbidity, expense and burden. This study may also identify previously unknown barriers to care that can be surmounted by innovative access and health care delivery approaches.

The primary objective is to evaluate an innovative approach for enhanced enrollment and engagement outreach intervention (EEE intervention) for rural veterans in VA health care services. This study entails a two-cell design, addressing this objective with a prospective, randomized controlled multi-site clinical trial that evaluates an active intervention compared to administrative outreach (AO, control condition) on whether or not a rurally-residing veteran obtains and attends a VA appointment.

DETAILED DESCRIPTION:
Access, enrollment, and engagement with primary and specialty health care services present significant challenges for rural populations worldwide. The Alabama Veterans Rural Health Initiative evaluated an innovative outreach intervention combining motivational interviewing, patient navigation, and health services education to promote utilization of the United States Veterans Administration Healthcare System (VA) by veterans who live in rural locations.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who live in rural Alabama counties who have either never enrolled or have previously enrolled but have not accessed a VA in 2 years or more
* Signed informed consent
* Any race, social class or ethnicity

Exclusion Criteria:

* Pending active legal charges or current/expected incarceration

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2010-10-01 (Actual); Study Completion 2013-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Davis, M.D., Principal Investigator — Tuscaloosa VAMC
Locations (2):
- United States (2):
  - Birmingham VAMC, Birmingham, Alabama
  - Tuscaloosa VAMC, Tuscaloosa, Alabama

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- [Result] Hilgeman MM, Mahaney-Price AF, Stanton MP, McNeal SF, Pettey KM, Tabb KD, Litaker MS, Parmelee P, Hamner K, Martin MY, Hawn MT, Kertesz SG, Davis LL; Alabama Veterans Rural Health Initiative (AVRHI) Steering Committee. Alabama Veterans Rural Health Initiative: a pilot study of enhanced community outreach in rural areas. J Rural Health. 2014 Spring;30(2):153-63. doi: 10.1111/jrh.12054. Epub 2013 Dec 15. PMID 24330220
- [Result] Mahaney-Price AF, Hilgeman MM, Davis LL, McNeal SF, Conner CM, Allen RS. Living will status and desire for living will help among rural Alabama veterans. Res Nurs Health. 2014 Oct;37(5):379-90. doi: 10.1002/nur.21617. Epub 2014 Aug 23. PMID 25156143
- [Result] Allen RS, Guadagno RE, Parmelee P, Minney JA, Hilgeman MM, Tabb KD, McNeil SF, Houston T, Kertesz S, Davis L. Internet connectivity among rural Alabama veterans: baseline findings from the Alabama Veterans Rural Health Initiative Project. Rural Remote Health. 2013 Apr-Jun;13(2):2138. Epub 2013 Jan 21. PMID 23331256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Rural veterans unlikely to be currently receiving VHA services were targeted for outreach, and therefore, recruitment design did not represent a population-based sampling strategy.
Groups:
- Enhanced Enrollment and Engagement (EEE): The EEE intervention includes 1) an educational video about the services and mission of the VHA to mitigate possible negative beliefs about the VHA system of care; 2) a motivational interviewing component to address ambivalence and promote behavior change; and 3) a patient navigator model to help patients overcome systems barriers to enrolling and obtaining an initial appointment. This intervention was provided by a rural health outreach worker.
- Administrative Outreach (AO): The Administrative Outreach (AO) includes a VHA enrollment document package without education, patient navigation, or motivational interview. The usual procedures for the VA to enroll the veteran were then followed by VA staff not associated with the research study.
Period: Overall Study
Arm/Group | Enhanced Enrollment and Engagement (EEE) | Administrative Outreach (AO)
Started | 101 | 102
Completed | 101 | 102
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Enhanced Enrollment and Engagement (EEE): The EEE intervention includes 1) an educational video about the services and mission of the VHA to mitigate possible negative beliefs about the VHA system of care; 2) a motivational interviewing component to address ambivalence and promote behavior change; and 3) a patient navigator model to help patients overcome systems barriers to enrolling and obtaining an initial appointment.
- Administrative Outreach (AO): The Administrative Outreach includes a VHA enrollment document package without education, patient navigation, or motivational interview. The usual procedures for the VA to enroll the veteran were then followed by VA staff not associated with the research study.
- Total: Total of all reporting groups
Arm/Group | Enhanced Enrollment and Engagement (EEE) | Administrative Outreach (AO) | Total
Number analyzed (Participants) | 101 | 102 | 203
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.72 (14.24) | 55.39 (14.60) | 55.6 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 95 | 94 | 189
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 49 | 34 | 83
  White | 52 | 67 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Attendance at a VA Appointment
Description: Attendance at a VA appointment was derived from VA clinical records, defined as the participant attending a scheduled VA clinic appointment. Participants who did not attend a VA clinic appointment be the end of 6-month observation period were classified as censored at 6 months.
Time Frame: 6 months
Population: Consenting participants who were randomized and lived in rural location.
Measure: Number; unit: participants
Groups:
- Enhanced Enrollment and Engagement(EEE): The EEE intervention includes 1) an educational video about the services and mission of the VHA to mitigate possible negative beliefs about the VHA system of care; 2) a motivational interviewing component to address ambivalence and promote behavior change; and 3) a patient navigator model to help patients overcome systems barriers to enrolling and obtaining an initial appointment.
Arm/Group | Enhanced Enrollment and Engagement(EEE) | Administrative Outreach (AO)
Number analyzed (Participants) | 101 | 102
participants | 88 | 59
Statistical Analysis 1: Comparison: Enhanced Enrollment and Engagement(EEE) vs Administrative Outreach (AO); Test type: Superiority; p < .0001, Chi-squared, Corrected

2. Secondary Outcome: Days Until VA Clinic Appointment
Description: The number of days from day of randomization to day that the participant attended the VA clinic appointment (derived from the VA medical records). Participants who did not attend a VA clinic appointment be the end of 6-month observation period were classified as censored at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Groups:
- Administrative Outreach (AO): Administrative Outreach (AO) includes a VHA enrollment document package without education, patient navigation, or motivational interview. The usual procedures for the VA to enroll the veteran were then followed by VA staff not associated with the research study.
Arm/Group | Enhanced Enrollment and Engagement (EEE) | Administrative Outreach (AO)
Number analyzed (Participants) | 101 | 102
days | 12 (49.8) | 98 (93.1)
Statistical Analysis 1: Comparison: Enhanced Enrollment and Engagement (EEE) vs Administrative Outreach (AO); Test type: Superiority; p < .0001, Log Rank; log rank Mantel Cox χ2 = 25.4

ADVERSE EVENTS:
Time Frame: 6 months
Description: same definition as clinicaltrials.gov
Groups:
- Enhanced Enrollment and Engagement (EEE): Enhanced Enrollment and Engagement (EEE) intervention includes 1) an educational video about the services and mission of the VHA to mitigate possible negative beliefs about the VHA system of care; 2) a motivational interviewing component to address ambivalence and promote behavior change; and 3) a patient navigator model to help patients overcome systems barriers to enrolling and obtaining an initial appointment.
Arm/Group | Enhanced Enrollment and Engagement (EEE) | Administrative Outreach (AO)
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/102
Serious Adverse Events (participants affected / at risk) | 1/101 | 2/102
Other Adverse Events (participants affected / at risk) | 0/101 | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Enrollment and Engagement (EEE) (N=101) | Administrative Outreach (AO) (N=102)
Hospitalization (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated hospitalization due to preexisting complication with pacemaker.
Death resulting from heart attack (Cardiac disorders) | 0 (0) | 1 (1) — Death unrelated to study procedures; a heart attack was reported as a cause of death, stemming from chronic heart disease
Hospitalization (Vascular disorders) | 0 (0) | 1 (1) — Hospitalization due to preexisting high blood pressure; not related to study procedures

LIMITATIONS AND CAVEATS:
Single geographic location; open label; bundled components of EEE intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No